CLINICAL TRIAL: NCT04946864
Title: A Phase Ib/II Study to Investigate the Safety, Tolerability, of APG-2575 as a Single Agent or in Combination With Systemic Anti-cancer Agents in Patients With ER Positive Breast Cancer or Advanced Solid Tumors.
Brief Title: A Study to Investigate the Safety, Tolerability, of APG-2575 as a Single Agent or in Combination for Breast Cancer
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG2575XU103
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Solid Tumor, Adult
MeSH Terms: conditions — Breast Neoplasms | interventions — Lisaftoclax; palbociclib

STUDY DESIGN:
Intervention Model Description: 3+3 cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- single arm (Experimental): APG2575
  Interventions: Drug: APG-2575
- combination arm (Experimental): APG2575+palbociclib i
  Interventions: Drug: APG-2575; Drug: Palbociclib

INTERVENTIONS:
Drug: APG-2575 — APG2575 monotherapy
  Other Names: APG2575
Drug: Palbociclib — combination APG2575+pablociclib
  Arms: combination arm

SUMMARY:
This is a multi-center, open-label, phase Ib/II study of APG-2575 as a single agent in patients with advanced solid tumors or in combination with anti-cancer agents such as CDK 4/6 inhibitor palbociclib in patients with ER+/HER2- metastatic breast cancer (mBC) who have progressed or relapsed after first line therapy

DETAILED DESCRIPTION:
The phase Ⅰb is dose escalation of APG-2575 as a single agent or in combination with palbociclib. A standard 3+3 design will be used to determine the MTD of APG-2575 as single agent in patients with solid tumors and MTD and RP2D of APG-2575 in combination with palbociclib in patients with breast cancer (MTD-combo). The phase II portion is a signal seeking expansion of APG-2575 at RP2D in combination with palbociclib in patients with ER+/HER2- metastatic breast cancers who have progressed during or relapsed after CDK 4/6inhibitor therapy. The phase Ⅱ portion will be conducted based on Simon's Minimax two stage design.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years. 2. Histologically or cytologically confirmed solid tumors; These locally advanced or metastatic diseases have no standard effective therapy available as judged by the investigator. 3. For the patients with breast cancer:

1. Must have histological or cytological confirmation of metastatic carcinoma of the breast (either from the primary or metastatic site), with the following tumor molecular characteristics (as determined from pre-screening testing):

   1. ER positive.
   2. HER2 negative - non-amplified (per ASCO/CAP guidelines).
2. Must have been treated with CDK4/6 inhibitor in the metastatic setting. And the patients must have experienced disease progression during or recurrence after CDK4/6 inhibitor therapy, which must have been administered for a minimum of 8 weeks prior to progression.
3. Must have measurable disease (according to RECIST v1.1) or evaluable disease. Boneonly metastases are allowed.
4. Physiological postmenopausal, defined as:

   1. Age ≥60 years, or
   2. Age <60 years and undergone bilateral oophorectomy or medically confirmed ovarian failure, or
   3. Age <60 years and have cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause and have serum levels of estradiol and FSH within the reference range for postmenopausal females.
   4. Premenopausal treated with LHRH analogues APG2575XU103 Version 1.0. / March 8, 2021 APG-2575 Ascentage Pharma Group Inc. Confidential Page 51 of 108 4. ECOG ≤ 1. 5. Adequate organ and bone marrow function within 14 days prior to registration:

1) Hemoglobin ≥ 90 g/L. 2) Absolute neutrophil count ≥ 1.5 x 109

* L. Note: Use of growth-factors to maintain ANC criterion is not permitted 3) Platelet count ≥ 100 x 109
* L. Note: Use of transfusions or thrombopoietic agents to achieve baseline platelet count criterion is prohibited. 4) ALT and AST ≤ 3 x upper limit of normal (ULN), or ≤ 5 x ULN if liver metastases are present. 5) Total serum bilirubin ≤ 1.5 x ULN. Patient's with Gilbert's syndrome may have a total serum bilirubin > 1.5 x ULN. 6) Serum creatinine ≤ 1.5 x upper limit of normal (ULN); if serum creatinine is >1.5 X ULN, creatinine clearance must be ≥ 50 mL/min (Cockcroft-Gault). 6. Female patients with childbearing potential must have negative urine or serum pregnancy test within 14 days prior to registration. 7. Able to swallow whole tablets. 8. Willingness to use contraception that is deemed effective for the patients with child bearing potential (postmenopausal women must have been amenorrhea for at least 12 months to be considered of non-childbearing potential) and their partners throughout the treatment period and for at least three months following the last dose of study drug.

  9. Brain metastases with clinically controlled neurologic symptoms. 10. Able to sign written informed consent with willingness and ability to comply with study procedures and follow-up examination. 11. Patient assigned to combination therapy, must provide sufficient archival tumor lesion or willing to provide fresh biopsy if no archival tissue available and core or excisional biopsy of a tumor lesion where feasible. Patients cannot provide a fresh biopsy (e.g. inaccessible or patient safety concern) may be eligible upon agreement from the sponsor. -

Exclusion Criteria:

* Receive any anti-cancer therapy within 14 days prior to the first dose of study drug, including chemotherapy, radiation therapy, surgery, targeted therapy, steroid therapy, endocrine therapy or other investigational therapy with the exception of hormones for hypothyroidism or estrogen replacement therapy (ERT) for non-breast cancer patients, or has had tumor embolization. Patients must have a 5x half-lives wash out time period or 14 for small molecules or 28 days for biologics including IO agents, gene or cellular therapeutic agents, respectively.

These following therapies are permitted:

a. Bisphosphonate or denosumab therapy for patients with bone metastases. APG2575XU103 Version 1.0. / March 8, 2021 APG-2575 Ascentage Pharma Group Inc. Confidential Page 52 of 108 b. Ovarian suppression in pre- and peri-menopausal patients. c. Palliative radiotherapy. 2. Receive any following agents within 14 days prior to the first dose of study drugs:

1. Strong CYP3A inhibitors or inducers
2. Drugs that are known to prolong the QT interval. 3. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to < Grade 2, exception being clinically insignificant toxicities of prior chemo/radiation such as lymphocytopenia or electrolyte abnormalities. 4. Pregnant or lactating. 5. Have a major surgery within 28 days from study entry, or have had minor surgery within 7 days of study entry. 6. Active symptomatic pathogenic infection including fungal, bacterial and/or viral infection including, but not limited to, active human immunodeficiency virus (HIV) or viral hepatitis (B or C) or active COVID-19. (Patients that have received a COVID-19 vaccination will be considered as eligible for the study.) 7. Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry. Patients with a QTc ≥ 480 msec (based on the mean value of the triplicate ECGs), family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes 8. Prior use of a Bcl-2 inhibitor. 9. Any other condition or circumstance that would, in the opinion of the investigator, make the patient unsuitable for participation in the study. -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days
  assessment of DLT for single and combination arm

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Emory University Hospital, Atlanta, Georgia
  - Next Oncology, Austin, Texas
  - MD Anderson, Houston, Texas
  - Next Oncology, San Antonio, Texas
- China (3):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital Sun Yat-Sen University, Guangdong, Guangzhou
  - Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No